CLINICAL TRIAL: NCT04767503
Title: The Impact of Different Anesthetic Methods on the Interaction of Gut Microbiota and Metabolomics Following Hepatectomy
Brief Title: Anesthesia on Gut Microbiota and Metabolomics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 201912148MINB
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Hepatic Tumor Resection
Keywords: hepatectomy; microbiota; metabolomics; anesthetic
MeSH Terms: interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Maintence of anesthesia during the operation using target control infusion with propofol 1mg/ml with bispetral index(BIS) in the range 40-60.
  Interventions: Drug: Propofol
- Desflurane (Sham Comparator): Maintence of anesthesia during the operation using inhalational agent desflurane with 0.5 to 1.5 minimal alveolar concentration (MAC) with bispetral index(BIS) in the range 40-60.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Propofol — Maintence of anestheisa with propofol guided by the bispectral index in the range 40-60.
  Arms: Propofol
Drug: Desflurane — Maintence of anestheisa with desflurane guided by the bispectral index in the range 40-60.
  Arms: Desflurane

SUMMARY:
Hepatectomies are performed for the treatment of hepatic tumors and livingdonor liver transplantation. The success of liver resection relies on the remnant liver's ability to regenerate after major tissue loss. Despite appropriate liver remnant volume after resection ensures the liver's ability to regenerate, regeneration progresses at variable ratesin patients.

Many researches have established a relationship between the gut microbiome and patients with liver disease such as liver cirrhosis, alcoholic liver disease and obesity related liver diseases. These liver disorders are associated with bacterial overgrowth, dysbiosis, and increased intestinal permeability. However, the relationship between hepatectomy and microbiota has not been fully investigated.

The measurement of small-molecule metabolites has been an integral part of clinical practice including the familiar clinical standards like glucose and creatinine. Metabolomics, however, is able to measure all the metabolites at once. It is possible to get a far more comprehensive picture of what is happening to a patient's physiology or metabolism. Although gut microbiota has been shown to be related to liver disease and liver regeneration. Obtaining a more comprehensive analysis by identifying not only the microbial composition but also the metabolites will be more insightful.

Many routine perioperative aspects of surgical care can impact the state of the microbiome and therefore can impact clinical outcomes, like bowel preparation and antibiotics. Potential factors affecting the gut microbiota also include perioperative manipulation, stress released hormones, and opioids. Maintenance of proper anesthetic depth is beneficial to attenuate surgical stress. General anesthesia including volatile anesthetics and opioids, is associated with altered gut microbiota which might in turn affect liver regeneration. In this regard, perioperative care such as anesthesia, is one of the key points for the success of a liver resection. However, which anesthetic method is preferable regarding postoperative outcome or recovery is controversial.

In this study, the study population will include liver tumor resection and living donor hepatectomy. We aimed to 1) identify the relationship of hepatectomy and changes of gut microbiota and metabolomics. 2) investigate the impact of different anesthetic methods on the interaction of gut microbiota and metabolomics.

ELIGIBILITY:
Inclusion Criteria:

1. Expected to receive hepatic tumor resection in National Taiwan University Hospital, age between 20 and 75 years old.

Exclusion Criteria:

1. Previous use of antibiotics within four weeks.
2. Previous gastrointestinal surgery.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiota analysis | one month
  16S metagenomic sequence processing
Metabolomics | one month
  Changes of metabolites in serum measured by metabolomic mass spectrometry

SECONDARY OUTCOMES:
I-FEED scoring | one week
  I-FEED scoring system for postoperative gastrointestinal function:
  1. Intake(score): tolerating oral diet(0), limited tolerance(1), complete Intolerance(3)
  2. Feeling nauseated(score): none(0), responsive to treatment(1), resistant to treatment(3)
  3. Emesis(score): none(0), ≧1 episode of low volume(<100mL) and none bilious(1), ≧1 episode of high volume(>100mL) or bilious(3)
  4. Exam(score): no distension(0), distension without tympany(1), significant distension with tympany(3)
  5. Duration of symptoms(score):0-24hours(0),24-72hours(1),>72hours(2)
  Total score: 0-2 normal, 3-5 postoperative GI intolerance, >6 postoperative GI dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Cheng Chan, M.D.,PhD., Principal Investigator — Department of Anesthesiology, National Taiwan University Hospital
Locations (1):
- Department of Anesthesiology, Taipei, Taiwan